CLINICAL TRIAL: NCT01444443
Title: DiaCon Closed-Loop Study
Brief Title: DiaCon Overnight Closed-Loop Glucose Control Study
Acronym: DiaCon2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Technical University of Denmark (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Signe Schmidt, MD, Clinical research fellow, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2106-07-0034
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Glucose control; Closed-loop; Insulin pump; Glucose sensor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-loop glucose control (Experimental): Blood glucose controlled by control algorithm.
  Interventions: Device: Closed-loop control
- Open-loop glucose control (Active Comparator): Blood glucose controlled by patient
  Interventions: Other: Open-loop control

INTERVENTIONS:
Device: Closed-loop control — Blood glucose controlled by algorithm
  Other Names: Metronic Veo-pump. DexCom 7+ sensor.
  Arms: Closed-loop glucose control
Other: Open-loop control — Blood glucose controlled by patient
  Arms: Open-loop glucose control

SUMMARY:
The objective of this in-clinic study is to test our closed-loop glucose control system in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Type 1 diabetes duration > 2 years
* HbA1c < 8%
* Insulin pump user > 1 year

Exclusion Criteria:

* Use of medication affecting glucose metabolism
* Pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic events | 22:00-07:00

SECONDARY OUTCOMES:
Time spent in euglycemia (3.9-8.0 mmol/l); mean blood glucose level; LBGI | 22:00-07:00

CONTACTS AND LOCATIONS:
Overall Officials: Signe Schmidt, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark